CLINICAL TRIAL: NCT00003115
Title: Spinal Effects of Epidural Hydromorphone
Brief Title: Epidural Hydromorphone Compared With Hydromorphone Infusion in Treating Patients With Prostate Cancer Undergoing Radical Prostatectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Dr. Oscar Deleon, Roswell Park Cancer Institute
Purpose: Supportive Care
Other Study IDs: CDR0000065866; RPCI-DS-95-35
Record Dates: First submitted 1999-11-01; First posted 2004-08-12 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Pain; Prostate Cancer
Keywords: prostate cancer; pain
MeSH Terms: conditions — Pain; Prostatic Neoplasms | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: hydromorphone hydrochloride

SUMMARY:
RATIONALE: Giving hydromorphone in different ways may relieve the pain associated with cancer surgery.

PURPOSE: Randomized double-blinded phase III trial to compare the effectiveness of epidural hydromorphone with hydromorphone infusion in patients with prostate cancer undergoing radical prostatectomy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Define the duration of action of hydromorphone (spinal vs supraspinal) in patients who have undergone radical prostatectomy. II. Demonstrate that the duration of the analgesic effects of equal blood concentrations of hydromorphone is dependent on the method used to attain this concentration by comparing continuous epidural infusion with that of a continuous intravenous infusion.

OUTLINE: This is a double blinded, randomized study. After all patients have undergone radical prostatectomy, hydromorphone is administered in two different ways. Patients receive either a hydromorphone bolus injection through an epidural catheter using a patient controlled analgesia pump or a hydromorphone bolus injection through an intravenous catheter using a patient controlled analgesia pump. Infusion for both groups is stopped at 24 hours. Patients are followed every 30 minutes for 6 hours.

PROJECTED ACCRUAL: A total of 40 patients will be accrued into this study over a 3 year period.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed prostate cancer Not metastatic Must be undergoing radical prostatectomy

PATIENT CHARACTERISTICS: Age: 18-70 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Neurologic: No presence of an intracranial lesion associated with increased intracranial pressure Pulmonary: No chronic obstructive pulmonary disease No cor pulmonale No emphysema No kyphoscoliosis No status asthmaticus Other: No contraindications for the insertion of epidural catheter No known hypersensitivity to hydromorphone No history of alcoholism, drug abuse, mental dysfunction, or cognitive deficiencies

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified for prior surgery(ies) Other: No preoperative opioids for any reason

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1996-06; Primary Completion 2003-01 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States